CLINICAL TRIAL: NCT03177902
Title: A Prospective Study to Assess Both Thyroid Abnormity Incidence In Chinese Women With Newly Diagnosed Breast Cancer and Thyroid Toxicity of Breast Cancer Patients Undergoing Chemotherapy
Brief Title: Evaluation of Thyroid Abnormity Incidence and Thyroid Toxicity During Chemotherapy Among Newly Diagnosed Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Qiong Wu, Principal Investigator, The First Affiliated Hospital of Bengbu Medical University
Other Study IDs: BYEC20170502
Record Dates: First submitted 2017-05-28; First posted 2017-06-06 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer Female; Thyroid Gland
MeSH Terms: conditions — Thyroid Diseases | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational group: Newly diagnosed breast cancer patients undergoing at least four cycles of chemotherapy
  Interventions: Drug: Chemotherapy
- Control group: Healthy Volunteers

INTERVENTIONS:
Drug: Chemotherapy — Newly diagnosed breast cancer patients undergoing at least four cycles of chemotherapy.
  Groups: Observational group

SUMMARY:
Breast cancer is one of the most common cancers in China. Even though advances in the field of breast cancer therapeutics, chemotherapy remains the mainstay therapeutic modality. The cytotoxic therapies are generally associated with some immediate or otherwise delayed side effects, such as adverse effects on gastrointestinal, hepatic, renal and hematological systems. The effect of chemotherapy on endocrine system, however, is comparatively less envisaged. Several epidemiological studies show a positive association between plasma thyroid hormones levels and breast cancer risk. Thyroid dysfunction is emerging as a variably common endocrine toxicity of several anticancer drugs. Due to the scarcity of data on the functioning of thyroid gland during chemotherapy in a large scale group, the present study was aimed to investigate the incidence of thyroid abnormity in Chinese women with newly diagnosed breast cancer, and also the effects of chemotherapy on thyroid gland functions or structure in these breast cancer patients undergoing at least four cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with histologically or cytologically proven primary breast cancer;
2. Age >18 years;
3. ECOG Performance Status: 0-2;
4. Life Expectancy: 3 months or more;
5. No previous anti-cancer therapy;
6. Be willing to undergo at least four cycles of anthracycline or taxane-based chemotherapy;
7. Adequate hematological, liver, and kidney functions.

Exclusion Criteria:

1. Pregnancy or lactation;
2. History of other malignancy or secondary breast cancer;
3. History of thyroid disease;
4. History of drug addiction or abuse;
5. History of immunodeficiency disease;
6. Treatment with drugs capable of influencing thyroid gland functions within 3 months prior to study entry;
7. Nonmeasurable disease such as un-controlled diabetes, severe cardiovascular and cerebrovascular diseases;
8. Current, recent (within 4 weeks prior to study entry), or planned participation in any other clinical trials;
9. Inability to understand and agree to informed consent.

Ages: 18 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed female breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-06-04 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants newly diagnosed with breast cancer | 1 week around the indicated detection point
  Rate of thyroid function (measured by chemiluminescence methods) or structure (measured by ultrasonic imaging) abnormity at the time of diagnosis and during chemotherapeutic period will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Wu, M.D.,Ph.D., Principal Investigator — First Affiliated Hospital of Bengbu Medical College
Locations (1):
- Department of Medical Oncology, First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China